CLINICAL TRIAL: NCT04733157
Title: The Efficacy of Tranexamic Acid in Preventing Postpartum Haemorrhage After Caesarean Section
Acronym: ETAPPH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Zimbabwe (Other)
Collaborators: Fogarty International Center of the National Institute of Health (NIH)
Responsible Party: Principal Investigator, Chipo Gwanzura, MD, Senior Registrar, University of Zimbabwe
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ETAPPH; D43TW009343 (NIH)
Record Dates: First submitted 2021-01-16; First posted 2021-02-01 (Actual); Results first posted 2023-03-20 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-02

CONDITIONS: Postpartum Hemorrhage
Keywords: Postpartum hemorrhage; Tranexamic acid; Caesarean section; Prevent
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Tranexamic Acid

STUDY DESIGN:
Intervention Model Description: This trial will be an open-label, two-centre, randomized control trial with two parallel groups including 1,162 women who undergo elective or emergency caesarean deliveries at term. The study group will receive TXA 1g intravenously at the onset of skin incision. There is normal saline placebo for the control group. The study and control groups will both receive the standard care offered at caesarean section including 5 IU of oxytocin intravenously on delivery of the baby.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Study group/Group A (Experimental): The study group will receive TXA 1g intravenously at the onset of skin incision.
  Interventions: Drug: Tranexamic acid injection
- Control group/Group B (Placebo Comparator): There is an equivalent volume of normal saline for the control group.
  Interventions: Other: Normal saline placebo

INTERVENTIONS:
Drug: Tranexamic acid injection — Tranexamic 1g administered intravenously at the onset of skin incision at caesarean section
  Other Names: TXA
  Arms: Study group/Group A
Other: Normal saline placebo — 10ml of normal saline will be administered intravenously at onset of skin incision at caesarean section to the placebo group
  Arms: Control group/Group B

SUMMARY:
This study seeks to determine if the using tranexamic acid prophylactically at caesarean section will prevent postpartum haemorrhage which is a major cause of maternal mortality in Zimbabwe and globally.

DETAILED DESCRIPTION:
This trial will be an placebo-controlled, two-centre, randomized control trial with two parallel groups including 1,162 women who undergo elective or emergency caesarean deliveries at term. The study group will receive tranexamic acid (TXA) 1g intravenously at the onset of skin incision. There is normal saline placebo for the control group. The study and control groups will both receive the standard care offered at caesarean section including 5 IU of oxytocin intravenously on delivery of the baby. .

ELIGIBILITY:
Inclusion Criteria: Women undergoing elective or emergency caesarean section with:

* Estimated gestational age of 37 weeks or more
* Live intrauterine foetus
* Elective or emergency caesarean delivery
* Signed informed consent

Exclusion Criteria:

* History of coagulopathies or conditions predisposing them to thromboembolic phenomena,
* seizure history,
* autoimmune disease,
* placental abruption,
* placenta praevia,
* abnormally adherent placentae if identified on prenatal ultrasound,
* eclampsia or HELLP syndrome,
* known hypersensitivity to TXA,
* planned general anaesthesia,
* caesarean delivery for the second twin or second/third triplet(s) after vaginal birth of the first twin,
* poor understanding of English/Shona languages,
* those who have received anticoagulants in the week before delivery
* persons-under-investigation for Coronavirus disease (COVID-19) and confirmed COVID-19 positive women

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1226 (Actual)
Dates: Start 2021-03-23 (Actual); Primary Completion 2021-12-14 (Actual); Study Completion 2021-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chipo Gwanzura, MD, Principal Investigator — University of Zimbabwe
Locations (2):
- Zimbabwe (2):
  - Parirenyatwa Group of Hospitals (Mbuya Nehanda Maternity Hospital), Harare
  - Sally Mugabe Central Hospital Maternity Unit, Harare

IPD SHARING:
Plan to Share IPD: No
It is not yet known if there will be a plan to make individual patient data (IPD) available.

REFERENCES:
- [Derived] Gwanzura C, Gavi S, Mangiza M, Moyo FV, Lohman MC, Nhemachena T, Chipato T. Effect of anesthesia administration method on apgar scores of infants born to women undergoing elective cesarean section. BMC Anesthesiol. 2023 Apr 27;23(1):142. doi: 10.1186/s12871-023-02098-w. PMID 37106343

RESULTS

PARTICIPANT FLOW:
Groups:
- Study Group/Group A_(Tranexamic Acid): The study group will receive TXA 1g intravenously at the onset of skin incision.
  Tranexamic acid injection: Tranexamic 1g administered intravenously at the onset of skin incision at caesarean section
- Control Group/Group B_(Placebo): There is an equivalent volume of normal saline for the control group.
  Normal saline placebo: 10ml of normal saline will be administered intravenously at onset of skin incision at caesarean section to the placebo group
Period: Overall Study
Arm/Group | Study Group/Group A_(Tranexamic Acid) | Control Group/Group B_(Placebo)
Started | 613 | 613
Completed | 611 | 613
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Study Group/Group A_(Tranexamic Acid) | Control Group/Group B_(Placebo) | Total
Number analyzed (Participants) | 611 | 613 | 1224
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.1 (6.2) | 28.3 (6.3) | 28.7 (6.3)
Age, Customized [Count of Participants; unit: Participants]
  Age Group: less than 18 years | 14 | 16 | 30
  Age Group: between 18-25 years | 168 | 195 | 363
  Age Group: between 26-35 years | 322 | 321 | 643
  Age Group: greater than 35 years | 107 | 81 | 188
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Females | 611 | 613 | 1224
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Weight (kg) [Mean (Standard Deviation); unit: kg] | 74.6 (16.2) | 73.5 (15.3) | 74.0 (15.8)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 29.5 (11.4) | 30.1 (19.6) | 29.8 (15.8)
Abnormal Placentation [Count of Participants; unit: Participants]
  No abnormal placentation | 1 | 0 | 1
  Abnormal placentation present | 610 | 613 | 1223
Anemia [Count of Participants; unit: Participants]
  Anemia | 29 | 20 | 49
  Not anemic | 582 | 593 | 1175
Comorbidities [Count of Participants; unit: Participants]
  Comorbidities present | 48 | 30 | 78
  No comorbidities | 563 | 583 | 1146
Fetal Macrosomia [Count of Participants; unit: Participants]
  Birth Weight <=4000g | 578 | 582 | 1160
  Birth Weight >4000g | 32 | 28 | 60
  Missing | 1 | 3 | 4
Gestational Age (Weeks) [Count of Participants; unit: Participants]
  37 Weeks | 93 | 76 | 169
  38 Weeks | 158 | 160 | 318
  39 Weeks | 147 | 139 | 286
  40 Weeks | 114 | 133 | 247
  41 Weeks | 60 | 64 | 124
  42+ Weeks | 39 | 41 | 80
History of PPH [Count of Participants; unit: Participants]
  has had PPH | 4 | 2 | 6
  No history of PPH | 603 | 608 | 1211
  Missing | 4 | 3 | 7
HIV status [Count of Participants; unit: Participants]
  HIV Positive | 62 | 59 | 121
  HIV Negative | 524 | 519 | 1043
  Unknown | 25 | 35 | 60
Multiple Pregnancy [Count of Participants; unit: Participants]
  Had Multiple Pregnancy | 41 | 20 | 61
  No Multiple Pregnancy | 570 | 593 | 1163
Number of Previous Cesarean Sections [Count of Participants; unit: Participants]
  None | 264 | 290 | 554
  One | 192 | 199 | 391
  Two | 127 | 104 | 231
  Three | 25 | 20 | 45
  Four | 3 | 0 | 3
Polyhydramnios [Count of Participants; unit: Participants]
  Polyhydramnios present | 2 | 1 | 3
  No polyhydramnios | 609 | 612 | 1221
Previous Surgery [Count of Participants; unit: Participants]
  had a previous surgery | 7 | 14 | 21
  No previous surgery | 604 | 599 | 1203
Uterine Fibroids [Count of Participants; unit: Participants]
  Uterine fibroids present | 7 | 5 | 12
  No uterine fibroids | 604 | 608 | 1212

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Postpartum Hemorrhage (PPH)
Description: Calculated estimated blood loss exceeding 1000ml. Estimated Blood Loss (EBL) was calculated using laboratory values of hemoglobin levels before and after procedure. Postpartum hemorrhage is defined as blood loss exceeding 1000mL after cesarean section.
Time Frame: Up to day 2 postpartum
Population: Postpartum hemorrhage defined as having a blood loss greater than or equal to 1000 mL using change in hemoglobin values. In the clinical trial, some participants in both arms had missing data because they did not have their laboratory measurements for hemoglobin done. In Group A (93 participants) and in Group B (87 participants) had missing assessments for PPH.
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group/Group A_(Tranexamic Acid) | Control Group/Group B_(Placebo)
Number analyzed (Participants) | 520 | 524
Participants
  Did not have PPH (blood loss <1000 mL) | 409 | 399
  Had PPH (blood loss >=1000 mL) | 111 | 125
Statistical Analysis 1: Comparison: Study Group/Group A_(Tranexamic Acid) vs Control Group/Group B_(Placebo); Test type: Other; p = 0.33, Chi-squared — Threshold for statistical significance was 0.05; Risk Ratio (RR) = 0.87, 95% CI 2-sided [0.69 to 1.09], Standard Error of Mean 0.1

2. Secondary Outcome: Blood Loss Using Hemoglobin Values
Description: Calculated blood loss using hemoglobin values. A mean value of blood loss calculated using hemoglobin values
Time Frame: Up to day 2 postpartum
Population: Average blood loss in mL calculated using laboratory hemoglobin values collected from participants before and after procedure.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Study Group/Group A_(Tranexamic Acid) | Control Group/Group B_(Placebo)
Number analyzed (Participants) | 513 | 516
mL | 537.2 (758.2) | 528.6 (1020.9)

3. Secondary Outcome: Mean Blood Loss as Estimated by Obstetrician
Description: Visually estimated blood loss at time of caesarean section. Attending obstetrician gave an estimated value of blood loss after delivery.
Time Frame: 2 hours
Population: Missing data for some participants due to estimates not being done at the time of delivery.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Study Group/Group A_(Tranexamic Acid) | Control Group/Group B_(Placebo)
Number analyzed (Participants) | 590 | 588
mL | 501.2 (209.8) | 495.0 (188.8)

4. Secondary Outcome: Occurrence of Postpartum Shock
Description: Number of participants who had hypovolemic shock related to PPH as determined by assessing BP and pulse.
Time Frame: Up to day 2 postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group/Group A_(Tranexamic Acid) | Control Group/Group B_(Placebo)
Number analyzed (Participants) | 611 | 613
Participants
  No postpartum shock | 603 | 611
  Postpartum shock | 8 | 2

5. Secondary Outcome: Use of Supplementary Uterotonic(s)
Description: Number of women requiring supplementary uterotonics
Time Frame: Up to day 2 postpartum
Population: Missing information about additional uterotonics for some participants due to data entry issues after delivery.
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group/Group A_(Tranexamic Acid) | Control Group/Group B_(Placebo)
Number analyzed (Participants) | 345 | 306
Participants
  No supplementary uterotonic | 93 | 74
  Supplementary uterotonic given | 252 | 232

6. Secondary Outcome: Postpartum Transfusion
Description: Number of women given postpartum transfusion
Time Frame: Up to day 2 postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group/Group A_(Tranexamic Acid) | Control Group/Group B_(Placebo)
Number analyzed (Participants) | 611 | 613
Participants
  transfusion given | 8 | 9
  no transfusion given | 603 | 604

7. Secondary Outcome: Emergency Surgery for PPH
Description: Number of participants who had emergency surgery for PPH including caesarean hysterectomies
Time Frame: Up to day 2 postpartum
Population: Missing information from some participants due to data entry issues.
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group/Group A_(Tranexamic Acid) | Control Group/Group B_(Placebo)
Number analyzed (Participants) | 607 | 605
Participants
  No emergency surgery | 603 | 601
  Emergency Surgery done | 4 | 4

8. Secondary Outcome: Change in Peripartum Haemoglobin
Description: Mean change in haemoglobin concentration between the study group, calculated hemoglobin values at day 2 postpartum minus baseline hemoglobin values.
Time Frame: Up to day 2 postpartum
Population: Missing values due to missing information if blood draws were not done within the required time frame.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Study Group/Group A_(Tranexamic Acid) | Control Group/Group B_(Placebo)
Number analyzed (Participants) | 555 | 567
g/dL | 1.1 (1.4) | 1.16 (1.7)

9. Secondary Outcome: Number of Participants With a Decrease in Peripartum Hemoglobin
Description: Number of participants with a drop in hemoglobin more than 2g/dL or less than 2g/dL
Time Frame: Up to day 2 postpartum
Population: Missing data a result of laboratory specimens not being collected at the expected time from participants
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group/Group A_(Tranexamic Acid) | Control Group/Group B_(Placebo)
Number analyzed (Participants) | 555 | 567
Participants
  drop less than 2g/dl | 438 | 442
  drop greater than or equal to 2g/dl | 117 | 125

10. Secondary Outcome: Change in Peripartum Haematocrit
Description: Mean change in haematocrit percentage between the study groups from baseline to day 2 postpartum
Time Frame: Up to day 2 postpartum
Population: Missing data due laboratory measurements not being done for some participants as samples were not taken within required time frame.
Measure: Mean (Standard Deviation); unit: percent of hematocrit change
Arm/Group | Study Group/Group A_(Tranexamic Acid) | Control Group/Group B_(Placebo)
Number analyzed (Participants) | 556 | 567
percent of hematocrit change | 3.8 (4.6) | 3.6 (4.6)

11. Secondary Outcome: Admission Into Intensive Care Unit
Description: Number of participants transferred to intensive care unit
Time Frame: Up to day 2 postpartum
Population: data entry error for missing participant data
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group/Group A_(Tranexamic Acid) | Control Group/Group B_(Placebo)
Number analyzed (Participants) | 600 | 606
Participants
  Admitted into intensive care unit | 75 | 75
  Not admitted to intensive care | 525 | 531

12. Secondary Outcome: Death From Any Cause
Description: Number of participants who died from any cause
Time Frame: Up to date of death or day 4 from admission
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group/Group A_(Tranexamic Acid) | Control Group/Group B_(Placebo)
Number analyzed (Participants) | 611 | 613
Participants
  Number of Participants who lived | 611 | 613
  Number of Participants who died | 0 | 0

13. Secondary Outcome: Blood Pressure Measurements
Description: Blood pressure at 15, 30, 45, 60, and 120 min after delivery
Time Frame: Up to 2 hours after the caesarean section
Population: Some participants did not have their systolic and diastolic blood pressure measurements done (missing data)
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Study Group/Group A_(Tranexamic Acid) | Control Group/Group B_(Placebo)
Number analyzed (Participants) | 609 | 610
mmHg
  systolic blood pressure 15 minutes after delivery | 132.2 (17.6) | 131.2 (18.0)
  diastolic blood pressure 15 minutes after delivery: number analyzed (Participants) | 607 | 608
  diastolic blood pressure 15 minutes after delivery | 64.9 (33.8) | 69.1 (62.3)
  systolic blood pressure 30 minutes after delivery: number analyzed (Participants) | 609 | 608
  systolic blood pressure 30 minutes after delivery | 118.3 (17.3) | 119.0 (16.5)
  diastolic blood pressure 30 minutes after delivery: number analyzed (Participants) | 591 | 586
  diastolic blood pressure 30 minutes after delivery | 61.8 (14.5) | 65.5 (40.3)
  systolic blood pressure 45 minutes after delivery: number analyzed (Participants) | 592 | 588
  systolic blood pressure 45 minutes after delivery | 117.8 (18.9) | 118.7 (18.3)
  diastolic blood pressure 45 minutes after delivery: number analyzed (Participants) | 602 | 608
  diastolic blood pressure 45 minutes after delivery | 69.2 (11.7) | 68.2 (12.8)
  systolic blood pressure 60 minutes after delivery: number analyzed (Participants) | 609 | 609
  systolic blood pressure 60 minutes after delivery | 123.6 (18.1) | 124.2 (16.2)

14. Secondary Outcome: Number of Mild Adverse Events
Description: Number of mild events of nausea, vomiting, sensation of rings or spots of light in the visual field, dizziness
Time Frame: Up to 24 hours after administration
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group/Group A_(Tranexamic Acid) | Control Group/Group B_(Placebo)
Number analyzed (Participants) | 611 | 613
Participants
  Nausea | 9 | 16
  No Nausea | 602 | 597
  Vomiting | 29 | 18
  No Vomiting | 582 | 595
  Dizziness | 12 | 14
  No Dizziness | 599 | 599

15. Secondary Outcome: Number of Severe Adverse Events
Description: * Deep vein thrombosis (if the diagnosis is confirmed by Doppler ultrasound)
  * Pulmonary embolism (if the diagnosis is confirmed by radiological examination)
  * Myocardial infarction
  * Seizure
  * Renal failure requiring dialysis
Time Frame: Up to day 3 postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group/Group A_(Tranexamic Acid) | Control Group/Group B_(Placebo)
Number analyzed (Participants) | 611 | 613
Participants
  Deep Vein Thrombosis | 0 | 0
  No Deep Vein Thrombosis | 611 | 613
  Pulmonary Embolism | 0 | 0
  No Pulmonary Embolism | 611 | 613
  Myocardial Infarction | 0 | 1
  No Myocardial Infarction | 611 | 612
  Seizures | 0 | 0
  No Seizures | 611 | 613
  Renal failure requiring dialysis | 0 | 0
  No Renal failure requiring dialysis | 611 | 613

16. Secondary Outcome: Any Other Unexpected Adverse Event
Description: Number of unexpected events during and after the adminstration of study drug and duration of observation
Time Frame: Up to day 3 postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group/Group A_(Tranexamic Acid) | Control Group/Group B_(Placebo)
Number analyzed (Participants) | 611 | 613
Participants
  Unexpected events | 0 | 0
  No unexpected events | 611 | 613

17. Secondary Outcome: Length of Hospital Stay
Description: Duration of hospital admission in days
Time Frame: Up to day 3 postpartum
Population: Missing data due to data entry errors
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Study Group/Group A_(Tranexamic Acid) | Control Group/Group B_(Placebo)
Number analyzed (Participants) | 603 | 605
days | 3.5 (1.1) | 3.5 (1.3)

ADVERSE EVENTS:
Time Frame: 1 week
Arm/Group | Study Group/Group A_(Tranexamic Acid) | Control Group/Group B_(Placebo)
All-Cause Mortality (participants affected / at risk) | 0/611 | 0/613
Serious Adverse Events (participants affected / at risk) | 0/611 | 1/613
Other Adverse Events (participants affected / at risk) | 50/611 | 48/613
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Group/Group A_(Tranexamic Acid) (N=611) | Control Group/Group B_(Placebo) (N=613)
Myocardial Infarction (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Group/Group A_(Tranexamic Acid) (N=611) | Control Group/Group B_(Placebo) (N=613)
Nausea (Gastrointestinal disorders) | 9 (9) | 16 (16)
Vomiting (Gastrointestinal disorders) | 29 (29) | 18 (18)
Dizziness (General disorders) | 12 (12) | 14 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-16): https://cdn.clinicaltrials.gov/large-docs/57/NCT04733157/Prot_SAP_000.pdf